CLINICAL TRIAL: NCT05308394
Title: Gut Permeability-related Inflammation and Cardiovascular Disease Risk in Normal-weight and Metabolically Healthy Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-22-28
Record Dates: First submitted 2022-03-11; First posted 2022-04-04 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators are collecting serum and fecal samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: The control group for this study will consist of individuals with normal BMI (18.5 - 24.9 kg/m2), body fat percent < 25% (male) or < 35% (female), and up to 1 other risk factor among the following: blood pressure > 130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, and HDL < 40 (male) or < 50 (female).
  Interventions: Other: No experimental intervention will take place - the study is cross-sectional. Each participant will provide biological samples.
- Normal-weight obesity: Individuals with normal-weight obesity will be defined as having normal BMI (18.5 - 24.9 kg/m2), body fat percent > 25% (male) or > 35% (female).
  Interventions: Other: No experimental intervention will take place - the study is cross-sectional. Each participant will provide biological samples.
- Metabolically Healthy Obesity: Metabolically healthy obesity will be defined as having an obese BMI (> 30 kg/m2), body fat percent < 25% (male) or < 35% (female), and up to 1 other risk factor among the following: blood pressure > 130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, and HDL < 40 (male) or < 50 (female).
  Interventions: Other: No experimental intervention will take place - the study is cross-sectional. Each participant will provide biological samples.
- Metabolic Syndrome: Metabolic syndrome will be defined using the international Diabetes Federation criteria of an obese BMI ( > 30 kg/m2) and 2 or more of the following risk factors: blood pressure > 130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, and HDL < 40 (male) or < 50 (female).
  Interventions: Other: No experimental intervention will take place - the study is cross-sectional. Each participant will provide biological samples.

INTERVENTIONS:
Other: No experimental intervention will take place - the study is cross-sectional. Each participant will provide biological samples. — Each participant will provide a blood and fecal sample.

SUMMARY:
The investigators are examining the extent gut permeability explains observed inflammation in normal-weight and metabolically healthy obesity (and potentially cardiovascular disease risk).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is responsible for 25% of deaths in the United States, and chronic inflammation contributes to risk. A growing body of evidence suggests that gut-derived bacterial components (e.g., lipopolysaccharide or LPS) entering the bloodstream when the gut barrier fails (i.e., intestinal permeability) are a prominent source of inflammation in cardiometabolic conditions such as metabolic syndrome, coronary artery disease, and type 2 diabetes. Two groups that are at > 2x the risk for CVD, but largely still free of overt disease, are those with metabolically healthy obesity and normal-weight obesity. Those with metabolically healthy obesity - defined as having an obese body mass index (BMI) but other clinical risk factors in the normal range (e.g., blood lipids) - and normal-weight obesity - defined as having a normal BMI yet high percent body fat - generally display little evidence of clinical risk, but present with elevated inflammatory markers including C-reactive protein (CRP), tumor necrosis factor (TNF)-a, and interleukin (IL)-6). Therefore, it is likely that chronic inflammation is largely driving CVD risk in metabolically healthy and normal-weight obesity, but the source of this inflammation remains unclear. The primary aim of the proposed project is to determine the extent that markers of intestinal permeability are elevated in metabolically healthy obesity and normal-weight obesity compared to healthy controls and individuals with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Control group: normal BMI, body fat percentage < 25% for men and < 35% for women, < 1 of the following: blood pressure >130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, HDL cholesterol < 40 mg/dL (men) or < 50 mg/dL (women).
* Normal-weight obesity group: normal BMI, body fat percentage > 25% for men and > 35% for women.
* Metabolically healthy obesity: BMI > 30, body fat percentage > 25% for men and > 35% for women, and < 1 of the following: blood pressure >130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, HDL cholesterol < 40 mg/dL (men) or < 50 mg/dL (women).
* Metabolic syndrome group: BMI > 30, body fat percentage > 25% for men and > 35% for women, and 2 or more of the following: blood pressure >130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, HDL cholesterol < 40 mg/dL (men) or < 50 mg/dL (women).

Exclusion Criteria:

* Presence of pacemaker
* Pregnant
* Cardiometabolic disease (e.g., diabetes, cardiovascular disease)
* Disease that is inflammatory in nature (e.g., inflammatory bowel disease, rheumatoid arthritis)
* Postmenopausal status
* Use of tobacco products
* Using illicit drugs
* Using lipid lowering drugs

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: The study populations of interest are those with normal weight obesity (normal BMI and high body fat percent) and metabolically healthy obesity (obese BMI, but largely normal cardiovascular risk factors).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Indicators of gut permeability | 1 year
  The investigators will measure serum markers of gut permeability as primary outcomes (i.e., lipopolysaccharide binding protein, soluble cluster of differentiation (CD)14, intestinal fatty acid binding protein).
C-reactive protein | 1 year
  The investigators will measure the marker of chronic inflammation C-reactive protein (CRP) using an ELISA.
Inflammatory cytokines | 1 year
  The investigators will measure a panel of serum inflammatory cytokines that includes granulocyte macrophage-colony stimulating factor (GM-CSF), interferon (IFN)-γ, interleukin (IL)-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-23, and tumor necrosis factor (TNF)-α using a bioplex assay.

SECONDARY OUTCOMES:
Fecal microbiota | 1 year
  The investigators will assess microbiota composition in a subset of individuals (~n=10 per group).

OTHER OUTCOMES:
Body composition assessment with dual-energy X-ray absorptiometry (DXA) | Through study completion, an average of 1 year
  The investigators will perform DXA scans on all participants to assess body composition parameters (i.e., body fat percent, lean mass, percent, visceral adipose tissue).
Lipid panel with Abbott Piccolo Xpress Clinical Chemistry Analyzer | Through study completion, an average of 1 year
  The investigators will perform a lipid panel on all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- 208 Nancy Randolph Davis, Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided